CLINICAL TRIAL: NCT04903717
Title: Pragmatic Trial Of Messaging to Providers About Treatment With Mineralocorticoid Receptor Antagonists
Brief Title: Pragmatic Trial Of Alerts for Use of Mineralocorticoid Receptor Antagonists
Acronym: PROMPT-MRA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: Vifor Pharma (Industry); Relypsa, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2000030513
Record Dates: First submitted 2021-05-21; First posted 2021-05-26 (Actual); Last update posted 2024-08-23 (Actual); Status verified 2024-08

CONDITIONS: Heart Failure With Reduced Ejection Fraction

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention - Best Practice Alert (Experimental): Providers randomized to the intervention arm will have a best practice alert appear for each of their eligible patients upon opening of the order entry screen in the patient's medical record which alerts to the presence of HFrEF and the fact that the patient is not currently prescribed an MRA. A link to an order set for MRAs (or to potassium binders should a patient be hyperkalemic) will provided, along with a link to current best practices surrounding the use of MRAs.
  Interventions: Behavioral: Best Practice Alert
- Usual Care (No Intervention): Providers will not receive a best practice alert for eligible patients and will continue to care for patients as usual.

INTERVENTIONS:
Behavioral: Best Practice Alert — Providers randomized to the intervention arm will have a best practice alert appear for each of their eligible patients upon opening of the order entry screen in the patient's medical record. This alert informs the provider to the presence of HFrEF and absence of MRA prescription, notes the patient's current LVEF, and notes the most recent labs, including NT-ProBNP, potassium, and creatinine. Providers will also have access to a link to best available guideline recommended information regarding use of MRAs and a link to both an order set for prescribing an MRA and an alternate order set with option for potassium monitoring should hyperkalemia be a concern. If a patient is hyperkalemic (i.e. K ≥ 5 mEq/L), a link to an order set for prescribing a potassium binder will be provided instead. If a provider feels that the recommended therapy is not indicated for a particular patient, he/she can select an available reason from the list provided within the alert.
  Arms: Intervention - Best Practice Alert

SUMMARY:
The primary objective of this study is to determine if a best practice alert (BPA) system that prompts providers to consider the addition of a mineralocorticoid receptor antagonist (MRA) in eligible patients with heart failure with reduced ejection fraction (HFrEF) will result in increased prescription of this guideline-recommended therapy. The system will also inform providers about FDA-approved potassium binders for the treatment of hyperkalemia if elevated potassium is a barrier for MRA use and will provide educational information on the evidence for MRA therapy in these patients.

DETAILED DESCRIPTION:
Despite the robust literature demonstrating improved outcomes with the use of mineralocorticoid antagonists (MRAs) in patients with heart failure with reduced ejection fraction (HFrEF), MRAs continue to be underused in clinical practice. This underuse often stems from the perceived risks of hyperkalemia, including a prior history of hyperkalemia and acute or chronic kidney disease, as well as the cautioned use for those with potassium greater than 5.0 mEq/L, as recommended in national societal guidelines. New potassium binders have recently been approved by the United States Food and Drug Administration (FDA) to treat hyperkalemia. It remains unknown if a best practice alert built into the clinical electronic health record can facilitate MRA prescription in eligible patients by providing guideline-based information about MRA recommendations and evidence, as well as informing practitioners about available treatments for hyperkalemia.

This is a pragmatic, cluster-randomized, open-label interventional trial to test the comparative effectiveness of an EHR BPA system that informs practitioners about MRAs for HFrEF and, if necessary, potassium-binders that are FDA-approved for hyperkalemia, versus usual care (no alert, current standard of care). One hundred and fifty outpatient Cardiology and Internal Medicine providers (to include physicians and advanced practice providers (nurse practitioners, physician assistants, and advanced practice registered nurses)) practicing at affiliated locations will be enrolled and undergo randomization to either the intervention (alert) group or a control (usual care) group. Those in the intervention group will receive an informational alert for their eligible adult outpatients (those with HFrEF not currently prescribed an MRA). Those in the control group will not receive any alerts and will continue to care for patients as usual. The primary outcome will be the proportion of patients with HFrEF who have an active prescription for an MRA at 6 months following randomization.

ELIGIBILITY:
Inclusion Criteria:

* Adults equal to or greater than 18 years of age
* Outpatients of providers randomized into the study within Internal Medicine and Cardiology outpatient clinics
* Diagnosis of heart failure with reduced ejection fraction (LVEF less than or equal to 40% on the most recent TTE)
* Registration in the Yale Heart Failure Registry (NCT04237701)
* Not currently prescribed an MRA

Exclusion Criteria:

* Absolute contraindication to MRAs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1210 (Actual)
Dates: Start 2021-11-03 (Actual); Primary Completion 2023-08-06 (Actual); Study Completion 2024-02-06 (Actual)

PRIMARY OUTCOMES:
Proportion of patients with an active prescription for an MRA | Measured at 6 months post-randomization
  Proportion of patients with an active prescription for an MRA, defined as a prescription present in the electronic health record for any drug in the MRA class that is active (not expired) and has remaining doses left at 6 months after the date of randomization.

SECONDARY OUTCOMES:
Number of MRA prescriptions | Within one year post randomization
  Number of any MRA prescription during study period.
Percentage of MRA prescriptions filled | Within 30 days of written prescription
  Percentage of prescriptions filled of initial MRA prescriptions written during the study period.
Time to first MRA prescription | From enrollment to time of MRA prescription
  Time (in days) to first MRA prescription
Percentage of patients with Hyperkalemia (K>5.0) | Within one year post randomization
  Percentage of patients experiencing hyperkalemia (K greater than or equal to 5.0 mEq/L)
Percentage of patients with Hyperkalemia (K>5.5) | Within one year post randomization
  Percentage of patients experiencing hyperkalemia (K greater than or equal to 5.5 mEq/L)
Percentage of patients with Hyperkalemia (K>5.0) with MRA | Within one year post randomization
  Percentage of patients experiencing hyperkalemia (K greater than or equal to 5.0 mEq/L) with an active MRA prescription
Percentage of patients with Hyperkalemia (K>5.5) with MRA | Within one year post randomization
  Percentage of patients experiencing hyperkalemia (K greater than or equal to 5.5 mEq/L) with an active MRA prescription
Percentage of patients with potassium binder prescription | Measured at 1 month post randomization
  Percentage of participants with active prescription for potassium binders
Percentage of patients with potassium binder prescription | Measured at 2 months post randomization
  Percentage of participants with active prescription for potassium binders
Percentage of patients with potassium binder prescription | Measured at 3 months post randomization
  Percentage of participants with active prescription for potassium binders
Percentage of patients with potassium binder prescription | Measured at 4 months post randomization
  Percentage of participants with active prescription for potassium binders
Percentage of patients with potassium binder prescription | Measured at 5 months post randomization
  Percentage of participants with active prescription for potassium binders
Percentage of patients with potassium binder prescription | Measured at 6 months post randomization
  Percentage of participants with active prescription for potassium binders
Percentage of patients with potassium binder + MRA prescription | Measured at 1 month post randomization
  Percentage of participants with active prescription for potassium binders and MRA
Percentage of patients with potassium binder + MRA prescription | Measured at 2 months post randomization
  Percentage of participants with active prescription for potassium binders and MRA
Percentage of patients with potassium binder + MRA prescription | Measured at 3 months post randomization
  Percentage of participants with active prescription for potassium binders and MRA
Percentage of patients with potassium binder + MRA prescription | Measured at 4 months post randomization
  Percentage of participants with active prescription for potassium binders and MRA
Percentage of patients with potassium binder + MRA prescription | Measured at 5 months post randomization
  Percentage of participants with active prescription for potassium binders and MRA
Percentage of patients with potassium binder + MRA prescription | Measured at 6 months post randomization
  Percentage of participants with active prescription for potassium binders and MRA
Type of potassium binder prescribed | First potassium binder prescribed at any point between enrollment and study completion
  Type of first potassium binder prescribed
Rationale for provider not prescribing an MRA if indicated (intervention group only) | Any rationale provided within one year post randomization
  Provider-documented (via the best practice alert) rationale for not prescribing indicated MRA (intervention group only)
Rationale for provider not prescribing a potassium binder if indicated (intervention group only) | Any rationale provided within one year post randomization
  Provider-documented (via the best practice alert) rationale for not prescribing indicated potassium binder (intervention group only)
Percentage of patients with ED visits | Measured at 1 month post randomization
  Percentage of patients with any ED visit
Percentage of patients with ED visits | Measured at 3 months post randomization
  Percentage of patients with any ED visit
Percentage of patients with ED visits | Measured at 6 months post randomization
  Percentage of patients with any ED visit
Percentage of patients with ED visits | Measured at 12 months post randomization
  Percentage of patients with any ED visit
ED visit count | Measured at 1 month post randomization
  Count of ED visits per patient
ED visit count | Measured at 3 months post randomization
  Count of ED visits per patient
ED visit count | Measured at 6 months post randomization
  Count of ED visits per patient
ED visit count | Measured at 12 months post randomization
  Count of ED visits per patient
Rates of Heart failure-related hospital admissions | Measured at 1 month post randomization
  Rates of HF-related hospital admissions (uses computations phenotype)
Rates of Heart failure-related hospital admissions | Measured at 3 months post randomization
  Rates of HF-related hospital admissions (uses computations phenotype)
Rates of Heart failure-related hospital admissions | Measured at 6 months post randomization
  Rates of HF-related hospital admissions (uses computations phenotype)
Rates of Heart failure-related hospital admissions | Measured at 12 months post randomization
  Rates of HF-related hospital admissions (uses computations phenotype)
Rates Outpatient visits | Measured at 1 monnh post randomization
  Rates of outpatient visits
Rate of Outpatient visits | Measured at 3 months post randomization
  Rates of outpatient visits
Rate of Outpatient visits | Measured at 6 months post randomization
  Rates of outpatient visits
Rate of Outpatient visits | Measured at 12 months post randomization
  Rates of outpatient visits
Rate of ED visit + IV diuretics | Measured at 1 month post randomization
  Rates of total ED visits in which a dose of IV diuretics was given
Rate of ED visit + IV diuretics | Measured at 3 months post randomization
  Rates of total ED visits in which a dose of IV diuretics was given
Rate of ED visit + IV diuretics | Measured at 6 months post randomization
  Rates of total ED visits in which a dose of IV diuretics was given
Rate of ED visit + IV diuretics | Measured at 12 months post randomization
  Rates of total ED visits in which a dose of IV diuretics was given
All-cause mortality | Measured at 1 month post randomization
  Rates of all-cause mortality
All-cause mortality | Measured at 3 months post randomization
  Rates of all-cause mortality
All-cause mortality | Measured at 6 months post randomization
  Rates of all-cause mortality
All-cause mortality | Measured at 12 months post randomization
  Rates of all-cause mortality
Total healthcare associated costs | Measured at 1 month post randomization
  Total healthcare-associated cost per patient
Total healthcare associated costs | Measured at 3 months post randomization
  Total healthcare-associated cost per patient
Total healthcare associated costs | Measured at 6 months post randomization
  Total healthcare-associated cost per patient
Total healthcare associated costs | Measured at 12 months post randomization
  Total healthcare-associated cost per patient
Rates of documented hyperkalemia at an ED visit | Within one year post randomization
  Documented hyperkalemia (K ≥ 5.5 mEq/L) at an ED visit
Rates of documented hyperkalemia at an outpatient visit | Within one year post randomization
  Documented hyperkalemia (K ≥ 5.5 mEq/L) at an outpatient visit
Rates of documented hyperkalemia during a hospital HF admission | Within one year post randomization
  Documented hyperkalemia (K ≥ 5.5 mEq/L) at an HF-related hospital admission
Frequency of outpatient potassium monitoring | Within one year post randomization
  Frequency of outpatient potassium monitoring
Frequency of outpatient potassium monitoring +/- MRA | Within one year post randomization
  Frequency of outpatient potassium monitoring for those with an active prescription of MRA vs. not
Frequency of outpatient potassium monitoring +/- potassium binder | Within one year post randomization
  Frequency of outpatient potassium monitoring for those with an active prescription of potassium binder vs. not

OTHER OUTCOMES:
Subgroup Analysis: Hyperkalemia at randomization | At randomization
  Hyperkalemia at randomization at both thresholds of ≥ 5.0 mEq/L and K ≥ 5.5 mEq/L
Subgroup Analysis: Prior hyperkalemia (IDC-10 Code) | From one year prior to randomization up to randomization
  Prior documentation of hyperkalemia by ICD-10 Code during the past 1 year
Subgroup Analysis: Prior hyperkalemia (K history) | From one year prior to randomization up to randomization
  Prior documentation of hyperkalemia by history of K 5.0 mEq/L during the past 1 year
Subgroup Analysis: Patient demographics | At randomization
  The following demographics subgroups will be captured: Age <65 years of age, sex, race
Subgroup Analysis: Chronic Kidney Disease | At randomization
  Chronic kidney disease (CKD) stage ≥ stage III, glomerular filtration rate (GFR) <60
Subgroup Analysis: Insurance status | At randomization
  Insurance status (commercial, public (Medicare, Medicaid), other, none)
Subgroup Analysis: GDMT medications | At randomization
  Number of concomitant active prescriptions for GDMT medications (beta blocker, ACEi/ARB/ARNI, SGLT2-inhibitor)
Subgroup Analysis: Provider type | At randomization
  The following provider characteristics will be captured: title (advanced practitioner, resident physician, fellow physician, attending physician), history of or current Cardiology fellowship training, years of training post-graduate medical school

CONTACTS AND LOCATIONS:
Overall Officials: Francis P Wilson, MD MSCE, Principal Investigator — Yale University
Locations (1):
- Cardiology/Internal Medicine Outpatient Clinics of Yale New Health System, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified data underlying results for publication will be shared upon publication.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Upon publication; indefinitely.

REFERENCES:
- [Derived] Clark KAA, Victoria-Castro AM, Ghazi L, Yamamoto Y, Coronel-Moreno C, Kadhim BA, Riello RJ 3rd, O'Connor K, Ahmad T, Wilson FP, Desai NR. Rationale, Design, and Patient Characteristics of a Cluster-Randomized Pragmatic Trial to Improve Mineralocorticoid Antagonist Use. JACC Heart Fail. 2024 Feb;12(2):322-332. doi: 10.1016/j.jchf.2023.08.025. Epub 2023 Nov 8. PMID 37943221